CLINICAL TRIAL: NCT00579475
Title: The Effect of Preoperative Treatment With Mifepristone on Uterine Fibroids and Breast Tissue
Brief Title: The Effect of Mifepristone on Uterine Fibroids and Breast Tissue
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Kristina Gemzell Danielsson, Professor, MD,PhD, Karolinska Institutet
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WMB300; MPA Dnr151:2003/4444
Record Dates: First submitted 2007-12-21; First posted 2007-12-24 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2007-12

CONDITIONS: Uterine Fibroids
Keywords: mifepristone; leiomyomas; breast epithelial cell proliferation
MeSH Terms: conditions — Leiomyoma | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- I (Active Comparator): Mifepristone (Mifegyne) 50 mg every other day for 3 months
  Interventions: Drug: Mifegyne

INTERVENTIONS:
Drug: Mifegyne — tablets, 50 mg every other day
  Arms: I
Drug: placebo
  Arms: Placebo

SUMMARY:
Uterine fibroids are a benign but common condition among women in reproductive age. It is one of the most common reasons for hysterectomy since it often causes bleeding problems sometimes leading to anemia. Several alternative treatment regimens have been investigated that could replace surgery. The antiprogesterone, mifepristone, is one of the most promising drugs that have been tested. In addition to the inhibiting effect on the growth of uterine fibroids antiprogestins have been proposed to have an antiproliferative effect on breast tissue.

The purpose of the present study is to evaluate the effect of mifepristone on the volume of uterine fibroids. The study will also address the effect of mifepristone on the breast tissue

DETAILED DESCRIPTION:
Other purposes of this study include:

* To develop a new non-surgical method for treatment of uterine fibroids
* To study the effect of mifepristone on the size of uterine fibroids
* To evaluate factors regulating fibroid growth by comparison with untreated fibroids and normal myometrium
* To study the effect of mifepristone on the amount of blood loss and pelvic pain in patients with fibroids
* To study the effect of mifepristone on proliferation of breast tissue

ELIGIBILITY:
Inclusion Criteria:

Uterine fibroids requiring treatment

* Good general health
* Willing and able to participate after giving informed consent

Exclusion Criteria:

* Need for immediate surgery
* Concomitant hormonal treatment (HRT)
* History of malignant disorder of the breast
* Any contraindication for mifepristone

Criteria for retrospective exclusion:

Subjects may be excluded from analysis if one of the following applies:

* Any violation of the study protocol
* Lack of essential data

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-11; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Myoma size | 2004 to 2007

SECONDARY OUTCOMES:
Breast epithelial cell proliferation | 2004 to 2007

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Gemzell Danielsson, Prof.MD.PHD, Principal Investigator — Karolinska Institutet
Locations (1):
- Dept of Obstetrics and Gynecology, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Berger C, Boggavarapu N, Norlin E, Queckborner S, Hornaeus K, Falk A, Engman M, Ramstrom M, Lalitkumar PGL, Gemzell-Danielsson K. Molecular characterization of PRM-associated endometrial changes, PAEC, following mifepristone treatment. Contraception. 2018 Oct;98(4):317-322. doi: 10.1016/j.contraception.2018.05.020. Epub 2018 Jun 8. PMID 29890128
- [Derived] Engman M, Varghese S, Lagerstedt Robinson K, Malmgren H, Hammarsjo A, Bystrom B, Lalitkumar PG, Gemzell-Danielsson K. GSTM1 gene expression correlates to leiomyoma volume regression in response to mifepristone treatment. PLoS One. 2013 Dec 4;8(12):e80114. doi: 10.1371/journal.pone.0080114. eCollection 2013. PMID 24324590
- [Derived] Engman M, Granberg S, Williams AR, Meng CX, Lalitkumar PG, Gemzell-Danielsson K. Mifepristone for treatment of uterine leiomyoma. A prospective randomized placebo controlled trial. Hum Reprod. 2009 Aug;24(8):1870-9. doi: 10.1093/humrep/dep100. Epub 2009 Apr 23. PMID 19389793
- [Derived] Engman M, Skoog L, Soderqvist G, Gemzell-Danielsson K. The effect of mifepristone on breast cell proliferation in premenopausal women evaluated through fine needle aspiration cytology. Hum Reprod. 2008 Sep;23(9):2072-9. doi: 10.1093/humrep/den228. Epub 2008 Jun 24. PMID 18579510